CLINICAL TRIAL: NCT00658983
Title: Autologous Platelet Enriched Gel Versus Metalloproteinase Inhibitor in the Healing of Chronic Lower Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Medtronic (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/049
Record Dates: First submitted 2008-04-07; First posted 2008-04-16 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Chronic Lower Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Autologous Platelet Enriched Gel
  Interventions: Other: Autologous Platelet Enriched Gel
- 2 (Active Comparator): Metalloproteinase Inhibitor (Promogran)
  Interventions: Other: Metalloproteinase Inhibitor

INTERVENTIONS:
Other: Autologous Platelet Enriched Gel — Treatment with Autologous Platelet Enriched Gel
  Arms: 1
Other: Metalloproteinase Inhibitor — Treatment with Metalloproteinase Inhibitor (Promogran)
  Arms: 2

SUMMARY:
Compare Autologous Platelet Enriched Gel versus Metalloproteinase Inhibitor in the healing of chronic lower leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* 18 year or older
* A non-healing chronic lower leg ulcer
* Platelet ranges of 150000 per ml circulating blood

Exclusion Criteria:

* Presence of a tumor or metastatic disease
* Hypersensitive to collagen regenerated cellulose
* Hemodynamic unstable patient
* Hypercoagulability
* Heart decompensation or angina pectoris

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-04-01 (Actual); Primary Completion 2010-08-20 (Actual); Study Completion 2010-08-20 (Actual)

PRIMARY OUTCOMES:
Wound healing | 6 weeks

SECONDARY OUTCOMES:
Wound healing | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Wim Bongaerts, MD, Principal Investigator — University Hospital, Ghent; Wouter De Moor, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be